CLINICAL TRIAL: NCT06950281
Title: Low Sodium Oxybate Use for Nocturnal Cluster Headache: Safety, Efficacy and Tolerability of JZP-258 (XYWAV) - a Phase 2 Randomized, Double-Blind, Placebo-Controlled, Bi-center Study.
Brief Title: Efficacy, Safety and Tolerability of Low Sodium Oxybate for Nocturnal Cluster Headache Attacks
Acronym: SUNCET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Rolf Fronczek, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136324
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Intervention Model Description: A 16 week, randomized, double-blind, placebo- controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum (Experimental): Low Sodium Oxybate (LXB) In this study we will use XYWAV, also known as JZP-258, oral solution 0.5 g/mL (Jazz Pharmaceuticals) for deepening sleep. JZP-258 is an oral solution containing LXB and is a central nervous system depressant. LXB will be administered as a twice nightly regimen. All subjects will undergo an 6 week Treatment Titration and Optimization Phase.
  Interventions: Drug: Low Sodium Oxybate
- Placebo (Placebo Comparator): Placebo will be administered as a twice nightly regimen. All subjects will undergo an 6 week Treatment Titration and Optimization Phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Sodium Oxybate — Low sodium oxybate (LXB) will be administered as a twice nightly regimen. All subjects will undergo an 6 week Treatment Titration and Optimization Phase. Titration should proceed in an increment of 1.5g per night each 7 days until a 50% reduction in nocturnal headache frequency is achieved or a maximum dose (9g per night) is reached. If a subject is unable to titrate to a higher dose, they may stay at the highest tolerated dose for the duration of the study. Subjects may stop titration or have dose reduction at any time for safety and tolerability reasons.
  Other Names: XYWAV; JZP-258
  Arms: Verum
Drug: Placebo — Placebo with equal appearance
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of low sodium oxybate (LXB) (brand name Xywav) in the treatment of (nocturnal) cluster headache attacks in subjects with chronic cluster headache.

It is an 16 week, randomized, double-blind, placebo- controlled, bi-center trial.

LXB will be administered as a twice nightly regimen. All subjects will undergo an 6 week Treatment Titration and Optimization Phase.

The main trial endpoint is the change from baseline in average weekly frequency of nocturnal cluster headache attacks over 4-week fixed stable dose of treatment period.

DETAILED DESCRIPTION:
The exact aetiology of cluster headache remains unknown and fundamental questions are still unanswered. However, the tendency of cluster headache attacks to occur during sleep suggests a pivotal role of the hypothalamus, a brain structure that regulates essential body functions such as sleep and the biological clock.

Low sodium oxybate (LXB) is a naturally occurring neurotransmitter and a psychoactive substance that deepens sleep by increasing slow wave sleep and reducing Rapid eye movement (REM) sleep. The chemical name of oxybate is gamma-hydroxybutyrate (GHB). The mechanism of action of LXB is still unknown. It is hypothesized that the therapeutic effects are mediated through GABA-B actions during sleep at noradrenergic and dopaminergic neurons, as well as at thalamocortical neurons.

We hypothesize that cluster headache attacks occur in relation to specific characteristics and time-points of the sleep microstructure and expect that a sleep-deepening treatment with LXB will reduce nocturnal attack-frequency and thereby improve sleep and quality of life.

The main objective of this study is to evaluate the efficacy and safety of LXB in the treatment of nocturnal cluster headache attacks in subjects with chronic cluster headache.

The main trial endpoint is the change from baseline in average weekly frequency of nocturnal cluster headache attacks over 4-week fixed stable dose of treatment period. Nocturnal attacks are defined as occurring after sleep onset during the night until morning awakening between 22:00 and 08:00.

Secondary endpoints include change from baseline in weekly frequency of cluster headache attacks in a 24-hr period (both nocturnal and day-time attacks) over 4-week fixed stable dose of treatment period. Additionally, the i) percentage of participants with a ≥50% reduction from baseline in the weekly number of nocturnal cluster headache attacks, ii) percentage of participants with a ≥50% reduction from baseline in the weekly number of cluster headache attacks in a 24-hr period (both nocturnal and day-time attacks) and iii) cluster headache attack pain intensity will be assessed over the 4-week fixed stable dose of treatment period, iv) Mean change in weekly number of times an abortive medication was taken v) number of patients with improvement in Patient Global Impressions Scale (PGIc) and Clinical Global Impressions Scale (CGIc) vi) improvement of sleep quality, sleep onset, sleep maintenance and sleep efficiency by diary. Optionally, two wearable skin sensors (Actiheart and CALERA Research) will be added for objective sleep and circadian rhythm measurements (including tri-axonal actigraphy, heart rate variability, core body temperature).

ELIGIBILITY:
Inclusion criteria

Age ≥18 and ≤75 at the time of consent.

Diagnosed with chronic cluster headache according to the International Classification of Headache Disorders (ICHD-III) criteria.

Free of other cluster headache prophylactic medication OR on stable dose for at least 4 weeks.

Not having received a GON (Greater Occipital Nerve) injection or oral prednisone in the previous 3 months.

At least 4 nocturnal cluster headache attacks per week (defined as occurring after sleep onset during the night between 22:00 and 08:00), not exclusively appearing during a single night, but spread across multiple nights.

Exclusion criteria

Suspected of having another trigeminal autonomic cephalalgia (TAC).

Other headaches if the patient cannot reliably distinguish them from cluster headache attacks.

Weight at inclusion of <50kg or >120kg.

Significant active or unstable psychiatric disease in the opinion of the investigator.

Significant pulmonary or neuromuscular diseases in the opinion of the investigator.

A history of or current indication of substance abuse or substance use disorder.

Unwillingness to refrain from consuming ≤ 1 alcohol unit per day and not later than 8 pm.

Stimulator devices which could influence sleep or cluster headache symptoms, such as an occipital nerve stimulator (ONS), when settings have not been stable for at least three months prior to screening.

Participation in a clinical trial of an investigation drug or device in the past 30 days.

Women who are pregnant/breastfeeding. Woman of childbearing age need to agree to sufficient contraception during the trial.

Contraindications for using LXB:

* Sleep apnoea syndrome or increased apnoea index (AI > 15/h).
* High risk of sleep apnoea syndrome, indicated by the STOP-Bang questionnaire (score ≥ 5).
* Currently suffering from severe depression and using medication or receiving cognitive therapy. Final choice is at the discretion of the principal investigator.
* Porphyria.
* Succinic semialdehyde dehydrogenase (SSADH-)deficiency.
* Use of opiates, barbiturates, valproic acid, phenytoin, ethosuximide, tricyclic antidepressants, topiramate, LXB (except for the intervention dose) or sedatives including benzodiazepines during the study. If benzodiazepines are used prior to inclusion, they must be discontinued at least one week before the baseline phase.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in average weekly frequency of nocturnal cluster headache attacks (verum vs placebo) | During 4-week fixed stable dose treatment phase
  During 4-week fixed stable dose treatment phase compared to baseline. Nocturnal attacks are defined as occurring after sleep onset during the night between 22:00 and 07:00. (verum vs placebo)

SECONDARY OUTCOMES:
Change in percentage of participants with a ≥30% reduction in the weekly number of nocturnal Cluster Headache Attacks | During 4-week fixed stable dose
  At week during 4-week fixed stable dose treatment phase compared to baseline.
Change in percentage of participants with a ≥50% reduction in the weekly number of nocturnal Cluster Headache Attacks | During 4-week fixed stable dose
  During 4-week fixed stable dose treatment phase compared to baseline.
Change in weekly frequency of cluster headache attacks in a 24-hr period during | During a 4-week fixed stable dose
  During a 4-week fixed stable dose treatment phase compared to baseline.
Change in percentage of participants with a ≥30% reduction in the weekly number of cluster headache attacks in a 24-hr period (daytime and nocturnal attacks) | During 4-week fixed stable dose
  During 4-week fixed stable dose treatment phase compared to baseline.
Change in percentage of participants with a ≥50% reduction in the weekly number of cluster headache attacks in a 24-hr period (daytime and nocturnal attacks) | During 4-week fixed stable dose
  During 4-week fixed stable dose treatment phase compared to baseline.
Change in pain scale (NRS 0-10) | During 4-week fixed stable dose
  During 4-week fixed stable dose treatment phase compared to baseline.